CLINICAL TRIAL: NCT01866137
Title: Copeptin During a Standardized Psychological Stress Test
Acronym: PsyCo
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: PsyCo
Record Dates: First submitted 2013-05-13; First posted 2013-05-31 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Stress
Keywords: Copeptin; psychological stress; The Trier Social Stress Test (TSST)
MeSH Terms: conditions — Diabetes Insipidus; Stress, Psychological

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 7.5 ml of EDTA blood, 7.5 ml of serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- no treatment: no treatment

SUMMARY:
The aim of the PsyCo Study is to determine whether psychological Stress has an influence on copeptin levels.

DETAILED DESCRIPTION:
healthy volunteers undergo the TSST and stress hormones as cortisol and copeptin are measured

ELIGIBILITY:
Inclusion Criteria:

•Aged over 18 years

Exclusion Criteria:

* Intake of any kind of medication (except birth control pill)
* BMI >30 kg/m2
* Evidence of any acute illness
* History of chronic illness
* Baseline glucose level >7 mmol/l Baseline sodium level <135 mmol/l or >145 mmol/l

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy adults
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-03; Primary Completion 2013-06 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Changes in copeptin levels after a psychological stress test in healthy volunteers | 30min before, at time point 0, +10, +20, +40, +60 after the psychological stress test

SECONDARY OUTCOMES:
Changes in copeptin levels after a psychological stress test in patients with central diabetes insipidus | Timpepoint 0, +10, +20, +40, +60 after the psychological stress test

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Christ-Crain, Prof.Dr.med., Principal Investigator
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland